CLINICAL TRIAL: NCT02727634
Title: Ultrapower, an In-house Developed System for Instantaneous Logging of Ultrasound Based Blood Flow, Blood Pressure and ECG.
Brief Title: Ultrapower; a Minimally Invasive Tool for Evaluation of Total Cardiac Power
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2016/49
Record Dates: First submitted 2016-03-17; First posted 2016-04-04 (Estimated); Last update posted 2019-03-27 (Actual); Status verified 2019-03

CONDITIONS: Cardiac Diseases
Keywords: Hemodynamics; Echocardiography, Doppler, Pulsed
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Postoperative elective CABG patients (Other): Patients included for coronary artery bypass graft (CABG) surgery, secondary to ischaemic heart disease.
  Interventions: Other: Comparison cardiac power and cardiac power output at different time points in the perioperative period

INTERVENTIONS:
Other: Comparison cardiac power and cardiac power output at different time points in the perioperative period — The intervention is a comparison between two methods of calculating the heart's energy delivery, cardiac power, measured in watts. A tertiary measurement is calculation of arterioventricular coupling. All patients will have cardiac power output calculated through the use of Doppler echocardiography. The echocardiography based cardiac output will be done through the velocity time integral of the left ventricular outflow tract (LVOT). This will be compared against total power as measured by our Ultrapower approach which involves instantaneous doppler measurement of cardiac output through LVOT multiplied with simultaneous radial artery pressure. This and ejection fraction (for calculation of ventriculoarterial coupling) will be recorded at rest in neutral position preoperatively, directly post operatively and the day after operation. Directly postoperatively the power measurements will also be repeated in Trendelenburg and anti Trendelenburg position.

SUMMARY:
The heart is essentially a hydraulic pump which ensures adequate delivery of blood through generating pressure and forward flow of blood. The energy delivered by the heart is uncommonly measured clinically, and todays gold standard involves placing a plastic catheter into the lung arteries. The investigators have developed an ultrasound based approach to calculate this energy without the need for catheters through the heart. This novel approach is called ultrapower. Ultrapower involves the instantaneous multiplication of the cardiac output and the arterial blood pressure. The study aims to use the ultrasound based approach to investigate Cardiac Power in the coronary artery bypass graft population.

ELIGIBILITY:
Inclusion Criteria:

• coronary artery bypass graft operation

Exclusion Criteria:

* Lack of informed consent
* Previous aortic valve replacement
* Inadequate Doppler signal on transthoracic echocardiography

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
The hearts energy delivery per second measured in watts (Cardiac Power), using two established methods and the ultrapower method | Immediately preoperatively
  Measured both as ultrapower and cardiac power output, both measured in watts and method of measurement described in intervention section
The hearts energy delivery per second measured in watts (Cardiac Power), using two established methods and the ultrapower method | approximately 1 hour post operatively
The hearts energy delivery per second measured in watts (Cardiac Power), using two established methods and the ultrapower method | 1 day after operation

CONTACTS AND LOCATIONS:
Overall Officials: Idar Kirkeby-Garstad, md phd, Principal Investigator — Norwegian University of Science and Technology
Locations (1):
- Department of cardiothoracic surgery, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: Undecided